CLINICAL TRIAL: NCT02996916
Title: Efficacy of Olmesartan on Cerebral Glucose Metabolism, Vascular Inflammation and Adipose Tissue
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kurume University (Other)
Responsible Party: Principal Investigator, Nobuhiro Tahara, Associate Professor, Kurume University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Olme-brain
Record Dates: First submitted 2016-12-13; First posted 2016-12-19 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Efficacy of Olmesartan on Cerebral Glucose Metabolism in Essential Hypertension
MeSH Terms: interventions — olmesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olmesartan (Active Comparator): Olmesartan 10-40mg daily
  Interventions: Drug: Olmesartan
- Amlodipine (Active Comparator): Amlodipine 2.5-10mg daily
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Olmesartan — 10-40mg daily
  Arms: Olmesartan
Drug: Amlodipine — 2.5-10mg daily
  Arms: Amlodipine

SUMMARY:
Hypertension is a leading risk factor for morbidity and mortality worldwide. The brain is a major target of the damaging effects of hypertension. Hypertension has been recognized as the leading cause of dementia as well as the most important risk factor for stroke and vascular cognitive impairment. Although glucose is the principal cerebral energy source, impact of hypertensive treatment on cerebral glucose metabolism is poorly understood.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Male and female subjects aged 20 years or older at informed consent
* Essential hypertension who had never received angiotensin II receptor antagonists and calcium channel blockers

Exclusion Criteria:

* Secondary hypertension or malignant hypertension
* Diabetes mellitus
* History or evidence of a stroke
* Hepatic or hematologic abnormality
* Mild Cognitive Impairment or Dementia
* Serum potassium level ≥ 5.5 mEq/L
* Serum creatinine level ≥ 3.0 mg/dL
* Acute or chronic disease
* Allergy to any drugs
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Effects of treatment on the nominal change in cerebral glucose metabolism from baseline after 6 months of treatment as measured by FDG-PET/CT | 6 months of treatment

SECONDARY OUTCOMES:
Change from baseline in vascular inflammation measured by blood-normalized standardized uptake value, known as a target-to-background ratio (TBR) by FDG-PET/CT | 6 months of treatment
Change from baseline in abdominal and muscle fat volume as measured by CT | 6 months of treatment
Change from baseline in circulating inflammatory markers including hsCRP (mg/L), adiponectin (µg/mL), ADMA (nmoL/mL), DPP-4 (ng/mL), advanced glycation end products (AGEs, µg/mL) and angiotensin-(1-7) (ng/mL) | 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhiro Tahara, MD, PhD, Study Chair — Department of Medicine, Division of Cardiovascular Medicine, Kurume University School of Medicine
Locations (1):
- Kurume University Hospital, Kurume, Japan

IPD SHARING:
Plan to Share IPD: Undecided